CLINICAL TRIAL: NCT00645606
Title: Single-agent Rituximab as Maintenance Treatment Versus Observation After Combined Induction Immunochemotherapy With Fludarabine, Cyclophosphamide and Rituximab in Patients Older Than 65 Years With Previously Untreated Chronic Lymphocytic Leukemia: a Phase III Trial of FILO
Brief Title: Rituximab Maintenance Versus Observation After First-line Immunochemotherapy by FCR in Older Patients With Chronic Lymphocytic Leukemia
Acronym: LLC2007SA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Roche Pharma AG (Industry); French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000589684; CHRUT-LLC-2007-SA (Other: CHU Tours); CHRUT-PHRN05-CD (Other: CHU Tours); INCA-RECF0497 (Other: INCA); 2007-001015-28 (EudraCT Number)
Record Dates: First submitted 2008-03-26; First posted 2008-03-27 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Leukemia
Keywords: B-cell chronic lymphocytic leukemia; Maintenance in first-line treatment; Elderly patients
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Observation (No Intervention): Observation every 8 weeks during 2 years
- rituximab arm (Experimental): rituximab :500 mg/m² every 8 weeks during 2 years
  Interventions: Biological: Rituximab

INTERVENTIONS:
Biological: Rituximab — rituximab :500 mg/m² every 8 weeks during 2 years
  Other Names: Mabthera
  Arms: rituximab arm

SUMMARY:
RATIONALE: Classical chemotherapy does not cure advanced chronic lymphocytic leukemia (CLL) despite new drugs. Rituximab is a monoclonal antibody directed against CD20 surface antigen on B lymphocytes and leads to apoptosis of CD20 positive B lymphocytes. The highest response rate yet published in the treatment of first-line CLL has been obtained by the association of fludarabine, cyclophosphamide and rituximab (FCR). Now, the question is whether this response can be improved, as some trials showed that eradication of minimal residual disease (MRD) in CLL is associated with a longer treatment-free and overall survival. Maintenance therapy using rituximab has been recently approved as a means of prolonging remission in patients with indolent non Hodgkin's lymphoma. Maintenance therapy with rituximab could be of interest in treatment of MRD in CLL and prolonging remission and survival times.

PURPOSE: The overall purpose of the study is to determine the value of immunotherapy maintenance with single agent rituximab in comparison with no further treatment (observation ) for previously untreated chronic lymphocytic leukaemia in elderly (>65 years) patients who respond to induction immunochemotherapy with FCR.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To demonstrate superiority, in terms of 3-year progression-free survival (PFS), of rituximab maintenance over observation in patients who are in complete or partial response (CR or PR) after induction therapy comprising fludarabine, cyclophosphamide, and rituximab.

Secondary

* To determine event-free survival, disease-free survival, overall survival, and time to next treatment, all from time of randomization.
* To determine overall response rate (CR and PR) according to NCI and iwCLL criteria
* To assess the rate of phenotypic response (minimal residual disease).
* To assess duration of phenotypic and NCI and iwCLL clinical responses.
* To determine response rates and time-related parameters in biological subgroups.
* To determine rates of treatment-related adverse events.
* To evaluate CD4/CD8 counts, immunoglobulin levels, and incidence of Coombs-positive hemolytic anemia.
* To study pharmacokinetics of rituximab during induction and maintenance.
* To evaluate the prognostic impact of the immunoglobulin FcγRIIIA genotype.
* To assess quality of life.
* To study pharmacoeconomics.

OUTLINE: This is a multicenter study. Randomization is stratified according to response to induction therapy (complete response [CR] vs partial response [PR]), IGHV mutational status, and 11q deletion.

Patients receive rituximab IV on days 1 and 14 of courses 1-2 and on day 1 of courses 3 and 4. Patients also receive oral fludarabine and oral cyclophosphamide once daily on days 2-4 of course 1 and on days 1-3 of courses 2-4. Courses are administered every 28 days. Patients achieving CR or PR are randomized 1:1 to maintenance arm or observation arm.

* Arm A: Patients receive rituximab IV every 2 months in the absence of disease progression or unacceptable toxicity for a maximum duration of 24 months (12 infusions).
* Arm B: Patients undergo observation only.

After completion of study therapy, patients are followed every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion criteria

* B-CLL
* Matutes score 4 or 5
* Binet stages B or C
* Age > 65 years old
* No previous treatment of CLL by chemotherapy, radiotherapy or immunotherapy, except glucocorticoids < 1 month
* Patient's written informed consent
* Life expectancy > 6 months

Exclusion criteria

* Binet stage A
* ECOG performance status 2 or more
* Presence of a 17p deletion by FISH (> 10% positive cores)
* Clinically significant auto-immune cytopenia, Coombs-positive hemolytic anemia as judged by the treating physician
* Patients with a history of another malignancy in complete remission less than 5 years, except basal cell skin cancer or tumor treated curatively by surgery
* Concomitant disease requiring prolonged use of corticosteroids (> 1 month)
* Any severe co-morbidities such as NYHA Class III or IV heart failure, myocardial infarction within 6 months, unstable angina, ventricular tachyarrhythmias requiring ongoing treatment, severe uncontrolled myocardiopathy, uncontrolled hypertension, severe chronic obstructive pulmonary disease with hypoxemia, or uncontrolled diabetes mellitus.
* CIRS (Cumulative Illness rating Scale) > 6
* Known hypersensitivity to murine proteins or to any of the study drugs or to their components
* Transformation into an aggressive B-cell malignancy (e.g. diffuse large cell lymphoma, Hodgkin lymphoma) or prolymphocytic leukemia
* Active bacterial, viral or fungal infection
* Seropositivity HIV, hepatitis C or hepatitis B (unless clearly due to vaccination)
* Total bilirubin, alkaline phosphatases and aminotransferases > 2 x ULN
* Creatinine clearance < 60 ml/min calculated according to the formula of Cockcroft and Gault
* Any coexisting medical or psychological condition that would preclude participation to the required study procedures
* Patient with mental deficiency preventing proper understanding of the requirements of treatment

Inclusion criteria at randomization

* Patients having received the full induction phase with 4 FC and 6 rituximab courses (with/without dose adjustments as per protocol)
* Complete or partial response according to NCI and iwCLL criteria at the end of induction phase
* Recovery from FCR toxicities
* Patient willingness to continue on protocol

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 542 (Actual)
Dates: Start 2007-12; Primary Completion 2014-02 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | randomization until disease progression or death
  Progression-free survival is defined as the time from randomization to the first occurrence of disease progression, relapse or death from any cause; using iwCLL criteria

SECONDARY OUTCOMES:
Event-free survival | randomization until disease progression, death, new CLL treatment, and secondary cancer
  Event-free survival is defined as the time from randomization to the occurrence of one of the following events, whichever occurs first: disease progression or relapse, death from any cause, initiation of any new anti-CLL therapy, and secondary malignancy
Disease-free survival | first documented CR until relapse
  Disease-free survival is defined as the time from first documented CR to relapse
Overall survival | randomization until death
  Overall survival is defined as the time from randomization to death from any cause
Time to next treatment | randomization until new CLL treatment
  Time to next treatment is defined as the time from randomization to initiation of a new CLL-related treatment
Overall response rate | baseline up to approximately 66 months
  Overall response rate is defined by the percentage of participants with an overall response; CR or PR according to NCI criteria and CR, CRi or PR according to iwCLL
Phenotypic response rate | randomization up to approximately 60 months
  Phenotypic response rate is defined by the percentage of participants with minimal residual disease negativity as measured by six-colour flow cytometry with a sensitivity of 0.7 x 10-5. MRD is considered as undetectable when the positivity criteria, defined as the presence of at least 20 CLL cells, is not reached
Rates of treatment-related adverse events | safety since baseline
  Rate of treatment-related adverse events (plus adverse events of particular interest) is defined as the percentage of participants with adverse events assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0 and version 2.0. for hematological toxicity
Pharmacokinetics of rituximab | baseline up to approximately 36 months
  Pharmacokinetics of rituximab during induction and rituximab maintenance
Quality of life | baseline up to approximately 30 months
  Change from baseline in EORTC Quality of Life Questionnaire Core 30

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Dartigeas, MD, Principal Investigator — Hématologie et Thérapie Cellulaire Hôpital Bretonneau CHU Tours FRANCE; Eric VAN DEN NESTE, MD PhD, Principal Investigator — Département d'hématologie Cliniques Universitaires Saint Luc BRUSSELS BELGIUM
Locations (1):
- French Innovative leukemia Organization, Tours, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dartigeas C, Van Den Neste E, Leger J, Maisonneuve H, Berthou C, Dilhuydy MS, De Guibert S, Lepretre S, Bene MC, Nguyen-Khac F, Letestu R, Cymbalista F, Rodon P, Aurran-Schleinitz T, Vilque JP, Tournilhac O, Mahe B, Laribi K, Michallet AS, Delmer A, Feugier P, Levy V, Delepine R, Colombat P, Leblond V; CLL 2007 SA investigators; French Innovative Leukemia Organization (FILO). Rituximab maintenance versus observation following abbreviated induction with chemoimmunotherapy in elderly patients with previously untreated chronic lymphocytic leukaemia (CLL 2007 SA): an open-label, randomised phase 3 study. Lancet Haematol. 2018 Feb;5(2):e82-e94. doi: 10.1016/S2352-3026(17)30235-1. Epub 2017 Dec 20. PMID 29275118